CLINICAL TRIAL: NCT06018948
Title: The Effect of Two Different Doses of Dexmedetomidine Infusion on Oxygenation, Lung Mechanics, and Quality of Recovery in Morbidly Obese Patients: A Prospective Randomized Controlled Study
Brief Title: Effect of Two Different Doses of Dexmedetomidine Infusion in Morbidly Obese Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Zeinab Tawfik, Assistant lecturer in Anesthesiology, Surgical ICU and Pain Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 33360/09/19
Record Dates: First submitted 2023-07-02; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anesthesia; Obesity, Morbid; Dexmedetomidine
MeSH Terms: conditions — Obesity, Morbid | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dexmedetomidine 0.6 group (Active Comparator): patients will receive a bolus dose of 1µg/kg dexmedetomidine15 minute after endotracheal intubation over 10 minutes followed by continuous infusion of 0.6 mic/kg/hour for one hour.
  Interventions: Drug: Dexmedetomidine 0.6
- Dexmedetomidine 0.3group (Active Comparator): patients will receive a bolus dose of 1µg/kg dexmedetomidine 15 minute after endotracheal intubation over 10 minutes followed by continuous infusion of 0.3 mic/kg/hour for one hour.
  Interventions: Drug: Dexmedetomidine 0.3
- Control group (Placebo Comparator): Patients will receive comparable volume of normal saline (0.9%) 15 minute after endotracheal intubation.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine 0.6 — Patients received a bolus dose of 1μg/kg Dexmedetomidine, 15 minutes after endotracheal intubation over 10 minutes followed by infusion of 0.6 μg/kg/hr for one hour.
  Arms: Dexmedetomidine 0.6 group
Drug: Dexmedetomidine 0.3 — Patients received a bolus dose of 1μg/kg Dexmedetomidine, 15 minutes after endotracheal intubation over 10 minutes followed by infusion of 0.3 μg/kg/hr for one hour.
  Arms: Dexmedetomidine 0.3group
Drug: Saline — Patients received over 10 minutes comparable volume of normal saline (0.9%) 15 min after endotracheal intubation followed by infusion.
  Arms: Control group

SUMMARY:
Compare the effects of two different doses of dexmedetomidine infusion on oxygenation as a primary outcome and on lung mechanics, quality of recovery and perioperative analgesia as secondary outcomes in morbidly obese patients with restrictive lung disease undergoing abdominal surgery.

DETAILED DESCRIPTION:
Dexmedetomidine is a selective α2 receptor agonist and has sympatholytic, analgesic, anti-inflammatory and sedative properties. Dexmedetomidine decreased dead space and improved both lung compliance and oxygenation in chronic obstructive pulmonary disease (COPD) patients undergoing lung cancer surgery.

The effects of dexmedetomidine on oxygenation and lung mechanics had been investigated in obstructive lung disease, but there are little information about its effect in morbidly obese patients with restrictive lung disease .

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index above 40 kg/m2 with restrictive lung disease((forced vital capacity) <70% in pre-operative pulmonary function tests), of American Society of anesthesiologists (ASA) physical status II and III.
* Aged 18-50 years.
* Scheduled for abdominal surgery.

Exclusion Criteria:

* Patients with Forced expiratory volume1/forced vital capacity<7.
* Uncontrolled cardiac, respiratory, hepatic or renal diseases.
* Allergy to the study drug

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Intraoperative oxygenation | Intraoperative
  Intraoperative oxygenation was assessed by P/F ratio (Arterial oxygen tension/fraction of inspired oxygen) at baseline and the end of drug infusion.

SECONDARY OUTCOMES:
Dynamic Lung compliance | Intraoperative
  Dynamic lung compliance=tidal volume/ (peak airway pressure- Positive end-expiratory pressure).
Post-operative pain | 24 hour postoperatively
  Assessment of post-operative pain by The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme
Dead space (dead space to tidal volume) | Intraoperative
  Physiological dead space was calculated by Hardman and Aitkenhead equation: (dead space to tidal volume) = 1.14(PaCO2 -EtCO2)/PaCO2- 0.005 dead space (%) = dead space by end of infusion - dead space at the base line / dead space by the end of drug infusion %
Quality of recovery score | 24 hours Postoperatively
  The Quality of recovery score scale provides a score ranging from 0 to 150, with a high score indicating a good quality of recovery
Time to first rescue analgesia | 24 hours Postoperatively
  Time to first rescue analgesia as morphine consumption was recorded
Static lung compliance | Intraoperative
  Static lung compliance =tidal volume /(plateau pressure - Positive end-expiratory pressure).
Lung compliance | 24 hours
  compliance = dynamic compliance at the end of the drug infusion - baseline dynamic compliance.
Plateau pressure | Intraoperative
  Plateau pressure was calculated by increasing end inspiratory pause to 30-40%.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: after the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author